CLINICAL TRIAL: NCT03616899
Title: A Phase 3, Double-masked, Randomized, Controlled Study of KPI-121 0.25% Ophthalmic Suspension Compared to Vehicle In Subjects With Dry Eye Disease (STRIDE 3)
Brief Title: Safety and Efficacy of KPI-121 in Subjects With DED
Acronym: STRIDE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-011
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-02

CONDITIONS: Kerato Conjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KPI-121 0.25% Ophthalmic Suspension (Active Comparator)
  Interventions: Drug: KPI-121 Ophthalmic Suspension
- Vehicle of KPI-121 0.25% Ophthalmic Suspension (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: KPI-121 Ophthalmic Suspension — KPI-121 Ophthalmic Suspension
  Arms: KPI-121 0.25% Ophthalmic Suspension
Drug: Vehicle — Vehicle for KPI-121 0.25% ophthalmic suspension
  Arms: Vehicle of KPI-121 0.25% Ophthalmic Suspension

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of KPI-121 0.25% ophthalmic suspension compared to vehicle (placebo) in subjects who have a documented clinical diagnosis of dry eye disease. The product will be studied over 14 days, with 1-2 drops instilled in each eye four times daily (QID).

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, double-masked, randomized, vehicle-controlled, parallel-group study designed to evaluate the safety and efficacy of KPI-121 0.25% ophthalmic suspension versus vehicle in subjects with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented clinical diagnosis of dry eye disease in both eyes

Exclusion Criteria:

* Known hypersensitivity or contraindication to the investigational product(s) or components
* History of glaucoma, IOP>21 mmHg at the screening or randomization visits, or being treated for glaucoma in either eye.
* Diagnosis of: ongoing ocular infection; severe/serious ocular condition that in judgment of Investigator could confound study assessments or limit compliance; or have been exposed to an investigational drug within 30 days prior to screening.
* In the opinion of the Investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (81):
- United States (81):
  - Investigator #133, Birmingham, Alabama
  - Investigator #278, Dothan, Alabama
  - Investigator #146, Chandler, Arizona
  - Investigator #148, Phoenix, Arizona
  - Investigator #280, Prescott, Arizona
  - Investigator #276, Sun City, Arizona
  - Investigator #185, Azusa, California
  - Investigator #143, Garden Grove, California
  - Investigator #147, Glendale, California
  - Investigator #272, Hemet, California
  - Investigator #155, Inglewood, California
  - Investigator #273, Long Beach, California
  - Investigator #130, Mission Hills, California
  - Investigator #247, Murrieta, California
  - Investigator #215, Newport Beach, California
  - Site #111, Rancho Cordova, California
  - Investigator #271, Santa Ana, California
  - Investigator #107, Torrance, California
  - Investigator #213, Westminster, California
  - Investigator #218, Littleton, Colorado
  - Investigator #184, Brooksville, Florida
  - Investigator #262, Delray Beach, Florida
  - Investigator #279, Fort Myers, Florida
  - Investigator #265, Jacksonville, Florida
  - Investigator #157, Largo, Florida
  - Investigator #189, Tampa, Florida
  - Investigator #136, Morrow, Georgia
  - Investigator #268, Roswell, Georgia
  - Investigator #266, Chicago, Illinois
  - Investigator #187, Hoffman Estates, Illinois
  - Investigator #151, Lake Villa, Illinois
  - Investigator #128, Indianapolis, Indiana
  - Investigator #250, Indianapolis, Indiana
  - Investigator #125, New Albany, Indiana
  - Investigator #274, Lexington, Kentucky
  - Investigator #195, Louisville, Kentucky
  - Investigator #168, Louisville, Kentucky
  - Investigator #219, Winchester, Massachusetts
  - Investigator #267, Kansas City, Missouri
  - Investigator #123, St Louis, Missouri
  - Investigator #106, St Louis, Missouri
  - Investigator #126, St Louis, Missouri
  - Investigator #131, Washington, Missouri
  - Investigator #281, Henderson, Nevada
  - Investigator #275, Las Vegas, Nevada
  - Investigator #263, Las Vegas, Nevada
  - Investigator #138, Las Vegas, Nevada
  - Investigator #105, New York, New York
  - Investigator #108, Rochester, New York
  - Investigator #132, Wantagh, New York
  - Investigator #264, Asheville, North Carolina
  - Investigator #217, Durham, North Carolina
  - Investigator #149, Durham, North Carolina
  - Investigator #102, High Point, North Carolina
  - Investigator #163, Raleigh, North Carolina
  - Investigator #282, Southern Pines, North Carolina
  - Investigator #269, Cincinnati, Ohio
  - Investigator #142, Cincinnati, Ohio
  - Investigator #137, Cleveland, Ohio
  - Investigator #171, Mason, Ohio
  - Investigator #224, Cranberry Township, Pennsylvania
  - Investigator #156, Kingston, Pennsylvania
  - Investigator #200, Lancaster, Pennsylvania
  - Investigator #277, West Mifflin, Pennsylvania
  - Investigator #240, Rapid City, South Dakota
  - Investigator #127, Memphis, Tennessee
  - Investigator #270, Austin, Texas
  - Investigator #188, Austin, Texas
  - Investigator #174, Cedar Park, Texas
  - Investigator #140, El Paso, Texas
  - Investigator #124, Houston, Texas
  - Investigator #259, Houston, Texas
  - Investigator #175, Lakeway, Texas
  - Investigator #182, League City, Texas
  - Investigator #191, League City, Texas
  - Site #177, San Antonio, Texas
  - Investigator #258, San Antonio, Texas
  - Investigator #186, San Antonio, Texas
  - Investigator #176, San Antonio, Texas
  - Investigator #222, Layton, Utah
  - Investigator #119, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 901 subjects were randomized and all were included in the ITT population.
Period: Overall Study
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Started | 447 | 454
Completed | 437 | 453
Not Completed | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension | Total
Number analyzed (Participants) | 447 | 454 | 901
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (15.26) | 57.3 (15.53) | 57.4 (15.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 330 | 669
  Male | 108 | 124 | 232
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 26 | 37 | 63
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 73 | 144
  White | 348 | 341 | 689
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 447 | 454 | 901

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline/Visit 2 (Day 1) in Ocular Discomfort Severity at Visit 4 (Day 15)
Description: Comparison of mean ocular discomfort severity between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: Intent to Treat population minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 434 | 451
score on a scale | -13.58 (19.379) | -8.91 (17.579)

2. Primary Outcome: Change From Baseline/Visit 2 (Day 1) Ocular Discomfort Severity at Visit 4 (Day 15) in the Subgroup of Participants With More Severe Ocular Discomfort
Description: Comparison of mean ocular discomfort severity between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse, in a sub-group of participants with more severe ocular discomfort at baseline.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: Sub-group of Intent to Treat population with more severe ocular discomfort minus subjects in each treatment group that discontinued the study by this time point or otherwise did not have this assessment completed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 296 | 304
score on a scale | -15.59 (20.373) | -10.15 (18.739)

3. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Bulbar Conjunctival Hyperemia at Visit 4 (Day 15)
Description: Comparison of mean bulbar conjunctival hyperemia between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-4 grading scale. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 432 | 449
score on a scale | -0.35 (0.575) | -0.18 (0.546)

4. Secondary Outcome: Change in Conjunctival Hyperemia Scores at Visit 4 (Day 15) by Alternate Assessor
Description: as for outcome 3
Time Frame: Baseline/Visit 2 (Day 1) and to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 437 | 453
score on a scale | -0.61 (0.646) | -0.48 (0.657)

5. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Ocular Discomfort Severity at Visit 3 (Day 8)
Description: as for outcome 1
Time Frame: Baseline/Visit 2 (Day 1) to Visit 3 (Day 8)
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 443 | 453
score on a scale | -8.05 (15.009) | -5.83 (15.176)

6. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Corneal Fluorescein Staining Score at Visit 4 (Day 15)
Description: Comparison of mean corneal fluorescein staining between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using methods developed by the National Eye Institute (NEI) Dry Eye Workshop in evaluating 5 regions of the cornea (superior, inferior, nasal, temporal and central) using a 0-3 grading scale, where 0 = no visible staining, 1 = Mild, 2 = moderate and 3 = severe.
Time Frame: Baseline/Visit 2 (Day 1) to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 437 | 453
score on a scale | -0.53 (0.800) | -0.43 (0.739)

7. Secondary Outcome: Change From Baseline/Visit 2 (Day 1) in Ocular Discomfort Severity at Visit 4 (Day 15) Using 7 Day Mean
Description: as for outcome 1
Time Frame: Baseline/Visit 2 (Day 1) to Visit 4 (Day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
Number analyzed (Participants) | 439 | 452
score on a scale | -11.76 (18.035) | -7.91 (16.298)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at Visit 2 (Day 1) until they exited the study at Visit 4 (Day 15).
Description: Subjects reported in each treatment arm come from the safety population and represent different numbers of subjects than that reported for efficacy (the ITT population). Two subjects Two subjects were randomized to vehicle (and were included in the vehicle arm for efficacy analyses as part of the ITT population) but erroneously received KPI-121 (and are therefore included in the KPI-121 treatment arm for safety analyses).
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle of KPI-121 0.25% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/449 | 0/452
Serious Adverse Events (participants affected / at risk) | 3/449 | 1/452
Other Adverse Events (participants affected / at risk) | 39/449 | 26/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 0.25% Ophthalmic Suspension (N=449) | Vehicle of KPI-121 0.25% Ophthalmic Suspension (N=452)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Delusional disorder, unspecified type (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 0.25% Ophthalmic Suspension (N=449) | Vehicle of KPI-121 0.25% Ophthalmic Suspension (N=452)
Eye irritation (Eye disorders) | 2 (3) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 3 (3)
Instillation site pain (General disorders) | 13 (13) | 7 (7)
Eye pruritus (Eye disorders) | 1 (1) | 3 (3)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Instillation site discharge (General disorders) | 1 (1) | 0 (0)
Instillation site pruritus (General disorders) | 1 (1) | 0 (0)
Corneal infiltrates (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 1 (1)
keratitis (Eye disorders) | 1 (1) | 0 (0)
Ocular hypaeremia (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Scleral hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1)
Conjunctival heamorrhage (Eye disorders) | 0 (0) | 1 (1)
Conjunctival vascular disorder (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eyelid pain (Eye disorders) | 0 (0) | 1 (1)
Eyelids pruritus (Eye disorders) | 0 (0) | 1 (1)
Growth of eyelashes (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Trichiasis (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreement between the Principal Investigator and the Sponsor restricts the PI's rights to discuss or publish trial results until after the first to occur of the following:

(a) publication of such multi-center clinical trial results; (b) notification by sponsor that such a multi-center clinical trial submission is no longer planned; or ( c) the eighteen ( 18) month anniversary of the completion, abandonment or termination of such multi-center clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT03616899/Prot_SAP_000.pdf